CLINICAL TRIAL: NCT03416075
Title: Risk Factors for Mortality in Patients With Interstitial Lung Disease Receiving Mechanical Ventilation: A Retrospective, Observational Cohort Study
Brief Title: Mechanical Ventilation in Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, Attending physician, Beijing Chao Yang Hospital
Other Study IDs: BeijingCYH-ICU-006
Record Dates: First submitted 2018-01-07; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Interstitial Lung Disease; Mechanical Ventilation; Risk Factors; Morality
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — Noninvasive and/or invasive mechanical ventilation were performed when patients had respiratory failure.

SUMMARY:
To identify risk factors for mortality in patients with interstitial lung disease receiving mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. They were clearly diagnosed as interstitial lung disease in hospital;
2. They had progressive worsening of dyspnea and their oxygenation indexes were less than 300 in ICU;
3. They received at least 48 hours of mechanical ventilation after being admitted into ICU.

Exclusion Criteria:

* We excluded patients who were admitted into ICU because of postoperative monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed as interstitial lung disease and received mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | 7 years

SECONDARY OUTCOMES:
Hospital mortality | 7 years
Noninvasive mechanical ventilation failure | 7 years
Invasive mechanical ventilation failure | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Zujin Luo, MD, Principal Investigator — Beijing Chao Yang Hospital

IPD SHARING:
Plan to Share IPD: No